CLINICAL TRIAL: NCT02373631
Title: Dry Needling Versus Conventional Physical Therapy in Patients With Knee Osteoarthritis: a Multi-center Randomized Clinical Trial
Brief Title: Dry Needling Versus Conventional Physical Therapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, DPT MSc FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0003
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling, Conventional PT (Experimental)
  Interventions: Other: Dry Needling, Conventional PT
- Conventional PT (Active Comparator)
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Dry Needling, Conventional PT — Dry needling to the knee and conventional physical therapy (stretching, ROM, strengthening), 1-2 treatments per week X6 weeks (up to 10 sessions total)
  Arms: Dry Needling, Conventional PT
Other: Conventional PT — Conventional physical therapy to include knee stretching, range of motion, and strengthening exercises,1-2 treatments per week X6 weeks (up to 10 sessions total)
  Arms: Conventional PT

SUMMARY:
The purpose of this research is to compare the effectiveness of conventional physical therapy (manual physical therapy, exercise, range of motion, and stretching) versus conventional physical therapy combined with dry needling in patients with knee osteoarthritis (OA). Physical therapists commonly use conventional physical therapy techniques and dry needling to treat knee OA, and this study is attempting to find out if the addition of dry needling to conventional physical therapy has an equal, greater, or lesser effect than conventional physical therapy alone.

DETAILED DESCRIPTION:
Patients with knee OA will be randomized to receive 1-2 treatments per week for 6 weeks (up to 10 sessions total) of either: (1) Dry Needling and conventional physical therapy or the (2) Conventional physical therapy (manual physical therapy, exercise, range of motion and stretching)

ELIGIBILITY:
Inclusion Criteria:

1. Report of knee pain of at least 2/10 per NPRS (0---10 scale) for >3 months
2. Report of at least 3 of the following per Altman et al. (1986)

   * Over 50 Years of age
   * Less than 30 minutes of morning stiffness
   * Crepitus on active motion
   * Bony tenderness
   * Bony enlargement
   * No palpable warmth of synovium

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: hypertension, infection, diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. History of previous surgery to the knee
3. History of physical therapy, massage therapy, chiropractic treatment, or injections for knee pain in the last 4 weeks
4. History of a surgical procedure on either lower extremity in last 6 months
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   * Weakness involving a major muscle group of the lower extremity.
   * Diminished patella or achilles tendon reflex
   * Diminished or absent sensation to pinprick in lower extremity dermatome
6. Involvement in litigation or worker's compensation regarding knee pain.
7. Any condition that might contraindicate the use of electro-needling
8. The patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity (NPRS) | Baseline, 2 Weeks, 6 Weeks, 3 Months
Change in Knee Osteoarthritis Index (Pain) | Baseline, 2 Weeks, 6 Weeks, 3 Months
  5 Questions each worth 0-4 points with a maximum score of 20 points possible
Change in Knee Osteoarthritis Index (Stiffness) | Baseline, 2 Weeks, 6 Weeks, 3 Months
  2 Questions each worth 0-4 points with a maximum score of 8 points possible
Change in Knee Osteoarthritis Index (Physical Function) | Baseline, 2 Weeks, 6 Weeks, 3 Months
  17 Questions each worth 0-4 points with a maximum score of 68 points possible
Change in Knee Osteoarthritis Index (Total) | Baseline, 2 Weeks, 6 Weeks, 3 Months
  24 Questions each worth 0-4 points with a maximum score of 96 points possible

SECONDARY OUTCOMES:
Change in Global Rating of Change Score (GROC) | 2 Weeks, 6 Weeks, 3 Months
Change in Medicine Intake (Frequency of medication intake) | Baseline, 3 months
  Frequency of medication intake (narcotics and over-the-counter) for knee pain

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT FAAOMPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States

REFERENCES:
- [Derived] Dunning J, Butts R, Young I, Mourad F, Galante V, Bliton P, Tanner M, Fernandez-de-Las-Penas C. Periosteal Electrical Dry Needling as an Adjunct to Exercise and Manual Therapy for Knee Osteoarthritis: A Multicenter Randomized Clinical Trial. Clin J Pain. 2018 Dec;34(12):1149-1158. doi: 10.1097/AJP.0000000000000634. PMID 29864043